CLINICAL TRIAL: NCT00749710
Title: Blood Loss and Complications of Internal Fixation of Femoral Neck Fractures in Patients Treated With Clopidogrel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Steinberg Ely MD, Tel-Aviv Sourasky Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-08-ES-143-CTIL; non
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2008-09-09 (Estimated); Status verified 2008-09

CONDITIONS: Femoral Neck Fractures; Pertrochanteric Fractures; Antiaggregant Therapy
Keywords: femoral neck fractures; pertrochanteric fractures; antiaggregant therapy; clopidogrel; plavix
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): immediate operation - ORIF - of hip fracture in patient treated with clopidogrel
  Interventions: Procedure: clopidogrel
- 2 (Active Comparator): ORIF - surgical treatment patients not on antiaggregant therapy
  Interventions: Procedure: no antiaggregant therapy

INTERVENTIONS:
Procedure: clopidogrel — ORIF - surgical treatment
  Arms: 1
Procedure: no antiaggregant therapy — ORIF - surgical treatment
  Arms: 2

SUMMARY:
Patients suffering from femoral neck or pertrochanteric fractures have a high rate of mortality and morbidity associated mainly with deconditioning and immobilization. Surgical management including open reduction and internaql fixation has been shown to reduce complication and improve outcome in such patients. Delay of surgery produces less optimal results and is associated with higher morbidity even after 24-48 hours of fracture event.

Patients treated with platelet antiaggregants are exposed to higher blood loss during surgery and related complications, as demonstrated in patients treated with Aspirin. However, cessation of antiaggregant therapy before surgery may be associated with complications of a hypercoagulable state and surgery delay.

Clpopidogrel is a fairly new approved antiaggregant drug indicated in cases of failed aspirin treatment in ischemic heart disease and cerebrovascular disease patients as well as in primary prevention of stent restenosis.

No data regarding complications of hip surgery in patients treated with Clpopidogrel is available.

Study hypothesis:

Definitive surgical treatment of patients treated with clopidogrel undergoing open reduction and internal fixation of pertrochnteric and femoral neck fractures is safe although associated with more extensive blood loss during surgery and postoperative wound complications.

ELIGIBILITY:
Inclusion Criteria:

* age > 60
* pertrochanteric or femoral neck fracture within 48 hours
* clopidogrel treatment - study group
* no antiaggregant treatment - control group
* ASA score <=3

Exclusion Criteria:

* hematologic malignancy
* hematologic malfunction
* warfarin treatment
* previous active GI or other internal bleeding - within 1 year
* thrombocytopenia < 150

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-09; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
mortality 30 days, 1 year functional score 1 year blood loss at surgery blood transfusions during hospitalization wound complications | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ely Steinberg, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center

REFERENCES:
- [Background] Wehren LE, Magaziner J. Hip fracture: risk factors and outcomes. Curr Osteoporos Rep. 2003 Sep;1(2):78-85. doi: 10.1007/s11914-003-0013-8. PMID 16036069